CLINICAL TRIAL: NCT05554575
Title: Safety and Efficacy of BT-007 CAR-T Cells in the Treatment of Patients With Relapsed/Refractory T Cell Lymphoblastic Lymphoma (R/R T-LBL)
Brief Title: Chimeric Antigen Receptor T-Cell (CAR-T) Cells in Patients With R/R T-LBL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioceltech Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-LBL-007-v2
Record Dates: First submitted 2022-09-13; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: T Cell Lymphoblastic Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BT-007 CD7 CAR-T cells in R/R T-LBL (Experimental): Subjects will receive BT-007 CD7 CAR-T cells infusion on Day 0 : 100% of total dose.
  Interventions: Biological: BT-007 CD7 CAR-T cells

INTERVENTIONS:
Biological: BT-007 CD7 CAR-T cells — T cells purified from the peripheral blood mononuclear cell (PBMC) of subjects or subjects' relatives which depend on their conditions, transduced with 4-1BB/CD3ζ lentiviral vector, expanded in vitro for future administration.

SUMMARY:
This is a single center, single arm, open-lable phase I study to determine the safety and efficacy of T cells expressing CD7 chimeric antigen receptors (referred to as "BT-007 CAR-T cells") in patients with relapsed or refractory acute T cell lymphoblastic lymphoma (R/R T-LBL).

DETAILED DESCRIPTION:
Primary objective:

To investigate the safety and efficacy of CD7 CAR-T cells in the treatment of patients with relapsed or refractory acute T cell lymphoblastic lymphoma (R/R T-LBL).

Secondary objective:

To assess the patient's quality of life after receiving the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD7 positive T-cell lymphoma confirmed by histology;
2. Relapsed refractory patients who received at least one line of systemic chemotherapy in the past;
3. At least one measurable target lesion;
4. Age: 18-70 years old (including 18 and 70 years old);
5. The expected survival period is more than 3 months;
6. Eastern Cooperative Oncology Group (ECOG) score 0-1;
7. Important organ functions met: left ventricular ejection fraction≥50% according to cardiac ultrasound; Serum Cr≤1.25 times the upper limit of normal range (ULN) or endogenous creatinine clearance≥45mL/min (Cockcroft Gault formula); ALT and AST≤3 times ULN, TBIL≤1.5 times ULN;
8. Blood routine: hemoglobin (Hgb)≥80g/L, neutrophil count (ANC)≥1×10^9/L, platelet PLT≥50×10^9/L；
9. Coagulation function: International standardized ratio (INR)≤1.5 times ULN; Activated partial thromboplastin time (APTT)≤1.5 times ULN (unless the subject is receiving anticoagulant treatment, and prothrombin time (PT)/INR and APTT are within the expected range of anticoagulant treatment at the time of screening);
10. The pregnancy test of women of childbearing age must be negative; Both male and female patients need to agree to use effective contraceptive measures during the treatment period and within the following 1 year;
11. Participate in this test voluntarily and sign the informed consent.

Exclusion Criteria:

1. Used immunosuppressive agents or therapeutic doses of corticosteroids (defined as prednisone>20mg or equivalent dose) within one week before blood collection, or used drugs that stimulate bone marrow hematopoiesis, such as Human Granulocyte Colony Stimulating Factor (G-CSF); But physiological substitution, topical or inhaled steroids are permitted;
2. Uncontrolled systemic active fungi, bacteria, viruses or other infections;
3. Active hepatitis B (HBV DNA>500IU/mL), hepatitis C (HCV RNA positive) or human immunodeficiency virus (HIV) antibody positive;
4. Central nervous system invasion, or central nervous system disease history, such as epilepsy, cerebrovascular disease, etc;
5. Pregnant or lactating women, or patients do not agree to use effective contraceptives during treatment and within the following 1 year;
6. Receiving allogeneic hematopoietic stem cell transplantation or organ transplantation;
7. Previous history of other malignant tumors. Patients with cured skin basal or squamous cell carcinoma and cervical carcinoma in situ at any time before the study were not included; Patients with other tumors not listed above, but which have been cured by surgery but not by other further treatment measures, and disease-free survival≥5 years, can be included in the study;
8. Patients with primary immunodeficiency or autoimmune diseases, but asymptomatic hypothyroidism, or well controlled type I diabetes can participate in this study;
9. Patients who participated in other clinical trials within 4 weeks before blood collection;
10. The investigator considers that there are other factors that are not suitable for inclusion or affect the subjects to participate in or complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | The changes between baseline and Day 28, Month 3, Month 6, as well as Month 24 for termination.
  The percentage of participants who achieved complete remission (CR) over all participants.
  The tumor status of patient is assessed for the baseline when assigned into treatment group. The overall CR is assessed by the Lugano Classification Lymphoma Response Criteria 2014 on Day 28, Month 3, Month 6, as well as Month 24 for termination. The overall CR is also assessed for the case withdraw from treatment before the termination of 24 months.
  The percentage of participants who achieved partial remission (PR) over all participants.
  The assessment criteria and time frame are the same as CR.

SECONDARY OUTCOMES:
The retention amount of CAR-T cells remaining in vivo | The retention amount of CAR-T cells in all subjects is assessed on Day 1, 7, 14, 28 during first month after cell infusion, and every month during Month 2 and 6, and every three months during Month 6 and 24 when terminated.
  The retention amount of CAR-T cells in all subjects within 24 months when terminated.
  The retention amount of CAR-T cells in all subjects is assessed on Day 1, 7, 14, 28 during first month after cell infusion. The retention amount is also assessed every month during Month 2 and 6, and every three months during Month 6 and 24 when terminated.
The retention time of CAR-T cells remaining in vivo | The retention time of CAR-T cells in all subjects is assessed on Day 1, 7, 14, 28 during first month after cell infusion, and every month during Month 2 and 6, and every three months during Month 6 and 24 when terminated.
  The retention time of CAR-T cells in all subjects within 24 months when terminated.
  The retention time of CAR-T cells in all subjects is assessed on Day 1, 7, 14, 28 during first month after cell infusion. The retention time is also assessed every month during Month 2 and 6, and every three months during Month 6 and 24 when terminated.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Liu, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided